CLINICAL TRIAL: NCT04822051
Title: The Effect of Psychoeducation Based On Uncertainty In Illness Theory On Intolerance To Uncertainty, Psychological Wellbeing And Coping Styles In Schizophrenia Caregivers
Brief Title: The Effect of Psychoeducation Based on Uncertainty In Illness Theory On Schizophrenia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sultan TAŞ BORA, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10386387
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Psychiatric Nursing; Schizophrenia
Keywords: caregiver; nursing theory; uncertainty in illness; psychoeducation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Masking Description: In this study, it is the same researcher who applied the intervention and evaluated the data.
  For this reason, a one-way blinding was made by ensuring that only the individuals who agreed to participate in the study did not know the group they were in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Group (Experimental): "Uncertainty Management Psychoeducation Program" was given.
  Interventions: Other: The Uncertainty Management Psychoeducation Program
- Control Group (No Intervention): No attempt was made by the researcher during the study. Only data collection was carried out.

INTERVENTIONS:
Other: The Uncertainty Management Psychoeducation Program — The program is conducted in the form of individual psychoeducation. The training was planned to include a total of five sessions, with 60 minutes for each session once a day, and at least two sessions a week. At least two days of a gap was decided between two consecutive sessions.
  Arms: Psychoeducation Group

SUMMARY:
The purpose of this study is to determine the effect of the psychoeducation program based on the Uncertainty in Illness Theory on intolerance to uncertainty, psychological well-being and coping styles of caregivers of schizophrenia patients.

Sample was 54 (experimental group:27; control group: 27) caregivers. Experimental group received psychoeducation program (5 sessions) based on Mishel's Reconceptualized Uncertainty in Illness Theory while control group did not receive any intervention. Data were collected 2 times: pre test, post test.

DETAILED DESCRIPTION:
It was determined that schizophrenia was seen in 19.78 million people in 2017 and constituted 0.51% of "disability adjusted life years" due to all causes. It has been determined that patients with schizophrenia have care needs in many areas related to daily care such as self-care, relationships and coping even in the early period after discharge. This situation shows that they need support to continue their daily life independently. In this context, families are the closest accessible support elements to the patients. Living with schizophrenia is a difficult situation to deal with for the family as well as for the patient. Caregivers in schizophrenia are dealing with an uncertain future accompanied by hope, fear, or both during the illness process.

Theorist Merle H. Mishel's Uncertainty in Illness Theory (UIT) emerged within the framework of the concept of "uncertainty in illness". The Reconceptualized Uncertainty in Illness Theory (RUIT) was developed to explain chronic conditions that cause individuals to experience uncertainty. "Uncertainty in illness" arises when disease-related processes have characteristics such as complexity, inconsistency, unpredictability, and lack of knowledge. RUIT provides a framework for nurses to develop interventions to improve psychological and behavioral outcomes that occur under uncertainty.Interventions for managing uncertainty help individuals gain knowledge, solve problems, see their health conditions manageable, and improve communication and coping skills. When RUIT based interventions are applied to cancer patients, many positive results have been reported in psychosocial aspects, especially in managing uncertainty.

This study that randomized controlled single blinded experimental nature, was conducted between April 2019 and August 2020 at psychiatry clinic with hospitalized schizophrenia patients caregivers, total of 54 including 27 interventions and 27 control groups. The data were collected by "Caregiver Information Form, Visual Analogue Scale, Intolerance to Uncertainty Scale, Psychological Well-being Scale, Stress Coping Styles Scale". The Uncertainty Management Psychoeducation Program, consisting of a total of five sessions was applied to the intervention group. No intervention was applied to the caregivers in the control group. The psychoeducational intervention, which was individually designed consisting of one session per day for each caregiver and five sessions with a gap of at least two days between sessions, was completed within two weeks. Pre-test and post-test measurements were also carried out during this period, and scales were applied for the pre-test at the beginning of the first session and for the post-test at the end of the last session. Mann-Whitney U and Wilcoxon tests were used for hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Being primarily responsible for the care of the patient diagnosed with schizophrenia according to The Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* For caregiver; being above 18 years of age
* Being literate
* For patient; being over 18 years of age
* Being diagnosed with schizophrenia for at least a year

Exclusion Criteria:

* Having any physical (hearing, speech, etc.) or mental disorder (psychotic disorder, mental retardation, etc.)
* Being a participant in a similar research
* For patient; having other accompanying mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Intolerance to uncertainty | 2 weeks
  Intolerance to Uncertainty Scale, consisting of 12 items. Intolerance to uncertainty is defined as "the tendency to react negatively to uncertain events and situations in cognitive, affective and behavioral terms Higher scores indicate a high level of intolerance to uncertainty. The highest score that can be obtained from the scale is 60 and the lowest score is 12.

SECONDARY OUTCOMES:
Perceived uncertainty | 2 weeks
  Visual analogue scale (VAS) is a scale used to convert some values that cannot be measured numerically into numerical ones. The two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line in the scale and one is asked to indicate where his condition is appropriate on this line. In the evaluation of the test, the values obtained for the individuals are averaged.
  VAS, was used to measure the level of uncertainty perceived by the individuals in this study. It is arranged in such a way that the level of uncertainty perceived by the caregiver can be marked on a ten-centimeter ruler with "no uncertainty" at the left end and "a high level of uncertainty" at the right. The lowest score that can be obtained from the scale is 0, the highest score is 10. 10 points indicates that the perceived level of uncertainty is too high.
Psychological well-being | 2 weeks
  Psychological Well-being Scale The scale has a single dimension and consists of 8 items. The items of the Psychological Well-Being Scale are answered between 1 and 7 as strongly disagree (1) and strongly agree (7). All items in the scale are expressed positively. Scores range from 8 (if all items are answered "strongly disagree") to 56 (if all items are answered "strongly agree"). A high score indicates that the person has psychological resources and strength.
Coping styles | 2 weeks
  Ways of Coping Questionnaire Scale measures two main styles of coping with stress. These are "Problem-oriented / active" and "Emotional / passive" styles. Higher scores obtained from self-confident, optimistic, and social support-seeking approaches mean that the person uses effective or active coping strategies, and higher scores from helpless and submissive approach scores mean that ineffective passive coping strategies are used. The scale is a 4-point Likert type consisting of 30 items and 5 separate subscales. Each item - totally unsuitable 0 points - unsuitable 1 point - suitable 2 points - totally appropriate 3 points. In the scale, the scores of each subscale are calculated separately and the total score for that subscale is obtained. 0-21 points for Self-Confident Approach, 0-24 points for Optimistic Approach, 0-15 points for the Social Support Seeking Approach, 0-12 points for Insecure Approach, 0-18 points for Submissive Approach.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Taş Bora, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not plan to share any data of participants.

REFERENCES:
- [Result] Bailey DE, Mishel MH, Belyea M, Stewart JL, Mohler J. Uncertainty intervention for watchful waiting in prostate cancer. Cancer Nurs. 2004 Sep-Oct;27(5):339-46. doi: 10.1097/00002820-200409000-00001. PMID 15525860
- [Result] Gil KM, Mishel MH, Belyea M, Germino B, Porter LS, Clayton M. Benefits of the uncertainty management intervention for African American and White older breast cancer survivors: 20-month outcomes. Int J Behav Med. 2006;13(4):286-94. doi: 10.1207/s15327558ijbm1304_3. PMID 17228986
- [Result] Mishel MH, Germino BB, Lin L, Pruthi RS, Wallen EM, Crandell J, Blyler D. Managing uncertainty about treatment decision making in early stage prostate cancer: a randomized clinical trial. Patient Educ Couns. 2009 Dec;77(3):349-59. doi: 10.1016/j.pec.2009.09.009. Epub 2009 Oct 9. PMID 19819096
- [Result] Germino BB, Mishel MH, Crandell J, Porter L, Blyler D, Jenerette C, Gil KM. Outcomes of an uncertainty management intervention in younger African American and Caucasian breast cancer survivors. Oncol Nurs Forum. 2013 Jan;40(1):82-92. doi: 10.1188/13.ONF.82-92. PMID 23269773
- [Result] Mishel MH, Belyea M, Germino BB, Stewart JL, Bailey DE Jr, Robertson C, Mohler J. Helping patients with localized prostate carcinoma manage uncertainty and treatment side effects: nurse-delivered psychoeducational intervention over the telephone. Cancer. 2002 Mar 15;94(6):1854-66. doi: 10.1002/cncr.10390. PMID 11920549
- [Result] Mishel MH. Uncertainty in illness. Image J Nurs Sch. 1988 Winter;20(4):225-32. doi: 10.1111/j.1547-5069.1988.tb00082.x. No abstract available. PMID 3203947
- [Result] Mishel MH. Reconceptualization of the uncertainty in illness theory. Image J Nurs Sch. 1990 Winter;22(4):256-62. doi: 10.1111/j.1547-5069.1990.tb00225.x. PMID 2292449
- [Result] Mishel MH, Germino BB, Gil KM, Belyea M, Laney IC, Stewart J, Porter L, Clayton M. Benefits from an uncertainty management intervention for African-American and Caucasian older long-term breast cancer survivors. Psychooncology. 2005 Nov;14(11):962-78. doi: 10.1002/pon.909. PMID 15712339
- [Result] Neville KL. Uncertainty in illness. An integrative review. Orthop Nurs. 2003 May-Jun;22(3):206-14. doi: 10.1097/00006416-200305000-00009. PMID 12803150
- [Result] He H, Liu Q, Li N, Guo L, Gao F, Bai L, Gao F, Lyu J. Trends in the incidence and DALYs of schizophrenia at the global, regional and national levels: results from the Global Burden of Disease Study 2017. Epidemiol Psychiatr Sci. 2020 Jan 13;29:e91. doi: 10.1017/S2045796019000891. PMID 31928566
- [Result] Taş S, Buldukoğlu K. Early period self-care ability and care requirements of schizophrenia patients after discharge. Journal of Psychiatric Nursing. 2018; 9(1):11-22.
- [Result] Williams LA. Theory of caregiving dynamics. In Smith MJ, Liehr PR, eds. Middle Range Theory for Nursing. New York: Springer Publishing Company; 2008.